CLINICAL TRIAL: NCT05471245
Title: AnGiographic Performance Following PCI With A Sirolimus-elutiNG Balloon in the TrEatment of De Novo CoronaRy Artery Disease: GINGER Study
Brief Title: AnGiographic Performance With A Sirolimus-elutiNG Balloon in the TrEatment of De Novo CoronaRy Artery Disease
Acronym: GINGER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Evidence per Attività e Ricerche Cardiovascolari ONLUS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GINGER
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Coronary Restenosis
Keywords: QCA; late loss; sirolimus eluting balloon
MeSH Terms: conditions — Coronary Restenosis

STUDY DESIGN:
Intervention Model Description: prospective enrolment of long lesions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- angiographic evaluation (Experimental): QCA at 9 months
  Interventions: Device: Magic Touch SCB by Concept Medical Inc.

INTERVENTIONS:
Device: Magic Touch SCB by Concept Medical Inc. — PCI with drug-coated balloon

SUMMARY:
Evaluate angiographic performance in long lesions of Sirolimus Eluting Balloon Magic Touch by Concept Medical

DETAILED DESCRIPTION:
To assess the angiographic performance of the Magic Touch Sirolimus-Coated Balloon (SCB) at 9 months follow-up after PCI for de novo CAD.

Primary end-points:

* Late lumen loss (LLL) at the SCB-treated segment within 9 months after the index procedure;
* Mean net lumen diameter gain at the SCB-treated segment at 9 months angiographic follow-up.

Secondary end-points:

* Procedural success defined as both SCB delivery and inflation at the "target" lesion site with <30% diameter stenosis (DS) in the SCB-treated segment and distal Thrombolysis In Myocardial Infarction (TIMI) 3 flow;
* Peri-procedural myocardial infarction (PMI) defined according to the EXCEL trial (creatinine kinase myocardial band) or Society for Cardiovascular Angiography and Interventions definitions (troponin);
* Binary restenosis rate at the SCB-treated segment at 9 months angiographic follow-up;
* A Device Oriented Composite End-point (DOCE) and its singular components (cardiac death, any target-vessel myocardial infarction excluding PMI, ischemia-driven target lesion revascularization) in-hospital, within 7 days after PCI; phone follow-up at 30-day (+/- 7 days) and 12 months (+/- 1 month) and a follow-up visit at 9 months (+/- 1 month). Any definite/probable SCB-treated segment thrombosis (in-hospital, within 7 days after PCI and at 30-day, 9-month, 1-year follow-up).

ELIGIBILITY:
Inclusion Criteria

1. Age >18 years
2. Patients presenting with stable or unstable coronary artery disease (CAD) eligible for percutaneous coronary intervention (PCI) with de novo CAD in one or two separates major epicardial territories and at least one lesion suitable for sirolimus coated balloon (SCB);
3. Reference vessel diameter (RVD) at the SCB target site ≥2.0 mm and ≤4.0 mm (by visual estimation and/or quantitative coronary angiography);
4. Lesion length at the SCB target site ≥25 mm;
5. Successful lesion preparation (full and homogenous pre-dilatation balloon expansion without type C-F dissection and/or TIMI flow=3 at the SCB target site;
6. SCB-target lesion located in the same or other vessels treated by drug-eluting stent (DES) implantation;
7. Patient able to understand and provide informed consent and comply with all study procedures including 9 months angiographic follow-up.

Exclusion criteria:

1. Patients participating in another clinical evaluation;
2. Age <18 years;
3. Cardiogenic shock;
4. Pregnancy or breastfeeding women; pregnancy test, either urine or blood test must be performed within 7 days prior to the index procedure in woman of child-bearing potential, and must not commit to initiating a pregnancy for 12 weeks after implantation, using effective contraception;
5. Thrombus containing lesion;
6. Unprotected left main as a target lesion unless this lesion is treated with a DES and SCB inflated distally or on a branch or on a different vessel;
7. Comorbidities with life expectancy <6 months;
8. Aorto-ostial target lesion (within 3 mm of the aorta junction); unless this lesion is treated with a DES and SCB inflated distally or on a branch or on a different vessel;
9. Target lesion located within an arterial or saphenous vein graft or distal to a diseased arterial or saphenous vein graft;
10. Every known allergy, intolerance or hypersensitivity to any medication used during the procedure and to drugs recommended after the procedure (e.g. aspirin, clopidogrel, ticagrelor, prasugrel);
11. Severe chronic kidney disease (glomerular filtration rate<30 ml/min/1.73 m2);
12. Platelet count <50,000cells/mm;
13. Stroke within the previous 6 months;
14. RVD at the SCB target site <2.0 mm or >4.0 mm (by visual estimation and/or QCA); target lesion with RVD larger than 4 mm can be treated with a DES and SCB inflated in other segments of the same or other vessels.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2025-10-08 (Actual); Study Completion 2025-10-08 (Actual)

PRIMARY OUTCOMES:
late lumen loss at 9 months measured by quantitative coronary angiography | 18 months
  QCA by core lab
incidence of adverse clinical events | 18 months
  myocardial infarction, death, need for revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Colombo, MD, Study Chair — Humanitas Research Hospital IRCCS, Rozzano-Milan
Locations (7):
- Italy (7):
  - IRCCS Ospedale San Raffaele, Milan, Italy/MI
  - Centro Cardiologico Monzino, Milan, Italy/MI
  - IRCCS Ospedale Galeazzi Sant'Ambrogio, Milan, Italy/MI
  - Istituto Clinico Humanitas, Rozzano, Italy/MI
  - Policlinico Universitario Campus Bio-Medico, Roma, Italy/RM
  - Policlinico Tor Vergata, Rome, Italy/RM
  - AULSS 2 Marca Trevigiana Ospedale di Conegliano, Conegliano, Italy/TV

IPD SHARING:
Plan to Share IPD: No
upon request

REFERENCES:
- [Background] Latib A, Colombo A, Castriota F, Micari A, Cremonesi A, De Felice F, Marchese A, Tespili M, Presbitero P, Sgueglia GA, Buffoli F, Tamburino C, Varbella F, Menozzi A. A randomized multicenter study comparing a paclitaxel drug-eluting balloon with a paclitaxel-eluting stent in small coronary vessels: the BELLO (Balloon Elution and Late Loss Optimization) study. J Am Coll Cardiol. 2012 Dec 18;60(24):2473-80. doi: 10.1016/j.jacc.2012.09.020. Epub 2012 Nov 14. PMID 23158530
- [Background] Tang Y, Qiao S, Su X, Chen Y, Jin Z, Chen H, Xu B, Kong X, Pang W, Liu Y, Yu Z, Li X, Li H, Zhao Y, Wang Y, Li W, Tian J, Guan C, Xu B, Gao R; RESTORE SVD China Investigators. Drug-Coated Balloon Versus Drug-Eluting Stent for Small-Vessel Disease: The RESTORE SVD China Randomized Trial. JACC Cardiovasc Interv. 2018 Dec 10;11(23):2381-2392. doi: 10.1016/j.jcin.2018.09.009. PMID 30522667
- [Background] Jeger RV, Farah A, Ohlow MA, Mangner N, Mobius-Winkler S, Weilenmann D, Wohrle J, Stachel G, Markovic S, Leibundgut G, Rickenbacher P, Osswald S, Cattaneo M, Gilgen N, Kaiser C, Scheller B; BASKET-SMALL 2 Investigators. Long-term efficacy and safety of drug-coated balloons versus drug-eluting stents for small coronary artery disease (BASKET-SMALL 2): 3-year follow-up of a randomised, non-inferiority trial. Lancet. 2020 Nov 7;396(10261):1504-1510. doi: 10.1016/S0140-6736(20)32173-5. Epub 2020 Oct 19. PMID 33091360
- [Background] Ono M, Kawashima H, Hara H, Katagiri Y, Takahashi K, Kogame N, Wykrzykowska JJ, Piek JJ, Doshi M, Sharif F, Onuma Y, Colombo A, Serruys PW, Cortese B. A Prospective Multicenter Randomized Trial to Assess the Effectiveness of the MagicTouch Sirolimus-Coated Balloon in Small Vessels: Rationale and Design of the TRANSFORM I Trial. Cardiovasc Revasc Med. 2021 Apr;25:29-35. doi: 10.1016/j.carrev.2020.10.004. Epub 2020 Oct 17. PMID 33109476
- [Background] Cortese B, Testa L, Di Palma G, Heang TM, Bossi I, Nuruddin AA, Ielasi A, Tespili M, Perez IS, Milazzo D, Benincasa S, Latib A, Cacucci M, Caiazzo G, Seresini G, Tomai F, Ocaranza R, Torres A, Perotto A, Bedogni F, Colombo A. Clinical performance of a novel sirolimus-coated balloon in coronary artery disease: EASTBOURNE registry. J Cardiovasc Med (Hagerstown). 2021 Feb 1;22(2):94-100. doi: 10.2459/JCM.0000000000001070. PMID 32740442
- [Background] Cortese B, Di Palma G, Latini R. Magic Touch(R): preliminary clinical evidence with a novel sirolimus drug coated balloon. Minerva Cardioangiol. 2018 Aug;66(4):508-517. doi: 10.23736/S0026-4725.18.04641-8. Epub 2018 Feb 19. PMID 29458247
- [Background] Stone GW, Sabik JF, Serruys PW, Simonton CA, Genereux P, Puskas J, Kandzari DE, Morice MC, Lembo N, Brown WM 3rd, Taggart DP, Banning A, Merkely B, Horkay F, Boonstra PW, van Boven AJ, Ungi I, Bogats G, Mansour S, Noiseux N, Sabate M, Pomar J, Hickey M, Gershlick A, Buszman P, Bochenek A, Schampaert E, Page P, Dressler O, Kosmidou I, Mehran R, Pocock SJ, Kappetein AP; EXCEL Trial Investigators. Everolimus-Eluting Stents or Bypass Surgery for Left Main Coronary Artery Disease. N Engl J Med. 2016 Dec 8;375(23):2223-2235. doi: 10.1056/NEJMoa1610227. Epub 2016 Oct 31. PMID 27797291
- [Background] Moussa ID, Klein LW, Shah B, Mehran R, Mack MJ, Brilakis ES, Reilly JP, Zoghbi G, Holper E, Stone GW. Consideration of a new definition of clinically relevant myocardial infarction after coronary revascularization: an expert consensus document from the Society for Cardiovascular Angiography and Interventions (SCAI). J Am Coll Cardiol. 2013 Oct 22;62(17):1563-70. doi: 10.1016/j.jacc.2013.08.720. PMID 24135581
- [Background] Garcia-Garcia HM, McFadden EP, Farb A, Mehran R, Stone GW, Spertus J, Onuma Y, Morel MA, van Es GA, Zuckerman B, Fearon WF, Taggart D, Kappetein AP, Krucoff MW, Vranckx P, Windecker S, Cutlip D, Serruys PW; Academic Research Consortium. Standardized End Point Definitions for Coronary Intervention Trials: The Academic Research Consortium-2 Consensus Document. Circulation. 2018 Jun 12;137(24):2635-2650. doi: 10.1161/CIRCULATIONAHA.117.029289. PMID 29891620
- [Background] Jeger RV, Eccleshall S, Wan Ahmad WA, Ge J, Poerner TC, Shin ES, Alfonso F, Latib A, Ong PJ, Rissanen TT, Saucedo J, Scheller B, Kleber FX; International DCB Consensus Group. Drug-Coated Balloons for Coronary Artery Disease: Third Report of the International DCB Consensus Group. JACC Cardiovasc Interv. 2020 Jun 22;13(12):1391-1402. doi: 10.1016/j.jcin.2020.02.043. Epub 2020 May 27. PMID 32473887
- [Background] Mehran R, Dangas G, Abizaid AS, Mintz GS, Lansky AJ, Satler LF, Pichard AD, Kent KM, Stone GW, Leon MB. Angiographic patterns of in-stent restenosis: classification and implications for long-term outcome. Circulation. 1999 Nov 2;100(18):1872-8. doi: 10.1161/01.cir.100.18.1872. PMID 10545431